CLINICAL TRIAL: NCT00024089
Title: A Phase II Study of ZD 1839 (Iressa) in Recurrent or Metastatic Squamous Cell Cancer of the Head and Neck
Brief Title: Gefitinib in Treating Patients With Recurrent and/or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068890; UUMC-8429-01; NCI-1701
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2005-11

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; salivary gland squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Gefitinib

ARMS (1):
- Arm I (Experimental): Patients receive oral gefitinib daily. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
Phase II trial to study the effectiveness of gefitinib in treating patients who have recurrent and/or metastatic head and neck cancer. Biological therapies such as gefitinib may interfere with the growth of tumor cells by blocking an enzyme necessary for cell growth.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the disease control rate, in terms of complete response, partial response, and stable disease for at least 4 months, in patients with recurrent and/or metastatic squamous cell cancer of the head and neck treated with gefitinib.

II. Determine the effect of this drug on epidermal growth factor receptor phosphorylation and expression of selected genes in these patients.

III. Determine the toxic effects of this drug in these patients.

OUTLINE: Patients are stratified as delineated in the Disease Characteristics.

Patients receive oral gefitinib daily. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary squamous cell cancer of the head and neck that is incurable by surgery or radiotherapy

  * Stratum I:

    * Failed surgery and/or radiotherapy and received no prior systemic chemotherapy for recurrent disease OR
    * Recurrent disease at least 6 months after prior multimodal primary therapy including neoadjuvant or concurrent chemotherapy OR
    * Metastatic disease at initial diagnosis and received no prior chemotherapy
  * Stratum II:

    * No more than 1 prior chemotherapy regimen for recurrent disease OR
    * Recurrent disease within 6 months after prior primary therapy that included chemotherapy
* Measurable disease

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Clear clinical evidence of progression or biopsy-proven residual cancer required if only site of measurable disease is in a previously irradiated field
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal (no greater than 1.5 times upper limit of normal [ULN] if liver metastases present)
* AST/ALT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No prior allergic reactions attributed to compounds of similar chemical or biologic composition to gefitinib
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior therapy with agents that target epidermal growth factor receptors

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy:

* No concurrent tamoxifen

Radiotherapy:

* Prior radiotherapy as primary or secondary treatment allowed
* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Prior surgery as primary or secondary treatment allowed
* At least 4 weeks since prior major surgery

Other:

* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV
* No concurrent 3A4 inhibitors (e.g., ketoconazole, erythromycin, verapamil)
* No concurrent drugs with known corneal toxicity (e.g., chlorpromazine, amiodarone, chloroquine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2001-07; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Disease control rate

SECONDARY OUTCOMES:
Biologic parameters
Toxicity
Response

CONTACTS AND LOCATIONS:
Overall Officials: Richard H. Wheeler, MD, Study Chair — University of Utah
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States